CLINICAL TRIAL: NCT03458234
Title: Pilot Study of Intra-Urethral Radiotransponder Beacon Guided Focal Prostate Stereotactic Body Radiotherapy
Brief Title: RAD 1801: Pilot Study of Intra-Urethral Radiotransponder Beacon Guided Focal Prostate Stereotactic Body Radiotherapy
Acronym: RAD1801
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer manufacturing radiotransponder beacons. No similar product available. The results are no longer expected to have a scholarly or clinical impact. Terminating the study before it reaches its target accrual.
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Andrew McDonald, Assistant Professor - Department of Radiation Oncology, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300002183; 000521070 (Other Grant/Funding Number: Varian Medical Systems)
Record Dates: First submitted 2018-03-01; First posted 2018-03-08 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
Keywords: Focal therapy; Prostate cancer; SBRT; Intra-urethral transponder
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Focal SBRT with intra-urethral radiotransponder (Experimental): This study will enroll patients that have a confirmed histology of prostate cancer. They will undergo a 3T MRI scan as well as a CT simulation with 16 French Foley Catheter containing dummy beacons for treatment planning purposes. The patient will then receive focal stereotactic body radiotherapy (SBRT) at a dose of 40 gy in 5 total fractions. Patients will be followed for 24 total months with specific follow-ups at 3, 6, 9, 12, 18, and 24 months.
  Interventions: Device: 16 French Foley Catheter

INTERVENTIONS:
Device: 16 French Foley Catheter — A Foley catheter is a medical apparatus that creates a passageway for the drainage and collection of urine. This type of catheter is made of a pliable material that indwells into an individual's bladder by way of the urethra.
  Featuring two separate channels down the tube, Foley catheters allow absolute stability and safe extraction. One channel of the catheter, by method of a balloon, is stabilized in a bladder; the other channel allows for the passage and collection of urine, by means of a leg bag or bedside drainage bag.
  Foley catheters are usually constructed out of either silicone or latex.

SUMMARY:
This study offers focal therapy for prostate cancer by using an intra-urethral radiotransponder temporarily placed during radiotherapy. The study aims to improve the risk-benefit ratio of therapy for early prostate cancer and potentially lessen symptom burden over time.

DETAILED DESCRIPTION:
This study offers focal stereotactic body radiotherapy for prostate cancer by using an intra-urethral radiotransponder placed temporarily during each of the 5 radiotherapy treatments. The study aims to improve the risk-benefit ratio of therapy for early prostate cancer and potentially lessen symptom burden over time while also accessing early efficacy, late toxicity, and overall quality of life post-treatment. Patients will be followed for 24 months (2 years) with follow-up appointments at 3, 6, 9, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically confirmed adenocarcinoma of the prostate, with biopsies obtained within 12 months of registration

  * Gleason score 3+3 or 3+4
  * PSA <10 ng/mL within 3 months of enrollment
  * Clinical stage T1a-T2a by digital rectal exam
  * Up to 2 intraprostatic nodules visible on MRI, with combined volume <50% of the total prostate volume
* Karnofsky Performance Status (KPS) >70%.
* Life expectancy >10 years
* Age ≥ 19 years
* Subjects given written informed consent

Exclusion Criteria:

* >2 MRI defined nodules representing prostate cancer
* Total volume of MRI nodules exceeding 50% of total prostate volume
* Positive biopsy core in sextant region without MRI defined nodule (i.e. biopsy proven MRI occult prostate cancer)
* American Urological Association (AUA) urinary score ≥ 18.
* History of inflammatory bowel disease.
* Prior pelvic surgery
* Prior treatment for prostate cancer
* Patients using immunosuppressive medications or other medications that may increase radiation toxicity such as methotrexate, sirolimus, tacrolimus, or colchicine that are unable to discontinue these medications during SBRT course. Use of corticosteroids is not considered an exclusion criteria.
* Platelet count < 70,000/µL
* Patients unable to discontinue anti-platelet or anti-coagulant medicine such as clopidogrel, dabigatran, warfarin, or low molecular weight heparin. Use of aspirin is not an exclusion criteria.
* Contraindication to MRI such as implanted devices.
* Metallic pelvic implants resulting in imaging artifact within the prostate on MRI or CT

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M McDonald, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Hazelrig-Salter Radiation Oncology Center, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Focal SBRT With Intra-urethral Radiotransponder: This study will enroll patients that have a confirmed histology of prostate cancer. They will undergo a 3T MRI scan as well as a CT simulation with 16 French Foley Catheter containing dummy beacons for treatment planning purposes. The patient will then receive focal stereotactic body radiotherapy (SBRT) at a dose of 40 gy in 5 total fractions. Patients will be followed for 24 total months with specific follow-ups at 3, 6, 9, 12, 18, and 24 months.
  16 French Foley Catheter: A Foley catheter is a medical apparatus that creates a passageway for the drainage and collection of urine. This type of catheter is made of a pliable material that indwells into an individual's bladder by way of the urethra.
  Featuring two separate channels down the tube, Foley catheters allow absolute stability and safe extraction. One channel of the catheter, by method of a balloon, is stabilized in a bladder; the other channel allows for the passage and collection of urine, by means of a leg bag or bedside drainage bag.
  Foley catheters are usually constructed out of either silicone or latex.
Period: Overall Study
Arm/Group | Focal SBRT With Intra-urethral Radiotransponder
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Focal SBRT With Intra-urethral Radiotransponder
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Confirm the Feasibility of Focal Prostate Stereotactic Body Radiotherapy (SBRT) With Real Time Guidance by Intra-urethral Radiotransponder Beacons.
Description: Confirm the technical feasibility of using focal prostate stereotactic body radiotherapy (SBRT) instead of traditional treatment methods using a 16-french Foley catheter and real time guidance by intra-urethral radiotransponder beacons.Feasibility will be defined as the ability of the treatment to take place as planned.
Time Frame: 2 years
Population: 5 patients signed consent, 1 patient withdrew consent prior to start of treatment. The funding source informed they are no longer manufacturing radiotransponder. No similar product. Therefore, no longer proceeding with study and no data collected.
Arm/Group | Focal SBRT With Intra-urethral Radiotransponder
Number analyzed (Participants) | 0

2. Secondary Outcome: Assess Early Efficacy
Description: Clinically assess early efficacy for men receiving focal prostate SBRT for low and low-intermediate risk prostate cancer.Efficacy will be defined as the absence of biochemically detected (via PSA lab testing) prostate cancer or clinically detected prostate cancer
Time Frame: Within 6 months of completion of radiation therapy
Population: as for outcome 1
Arm/Group | Focal SBRT With Intra-urethral Radiotransponder
Number analyzed (Participants) | 0

3. Secondary Outcome: Assess Late Toxicity
Description: Clinically assess late toxicity for men receiving focal prostate SBRT for low and low-intermediate risk prostate cancer. Late toxicity (defined as toxicity occurring >90 days after treatment) will be assessed with regular clinical exams and patient toxicity questionnaires.
Time Frame: Within 6 months of completion of radiation therapy
Population: as for outcome 1
Arm/Group | Focal SBRT With Intra-urethral Radiotransponder
Number analyzed (Participants) | 0

4. Secondary Outcome: Assess Quality of Life
Description: Clinically assess quality of life for men receiving focal prostate SBRT for low and low-intermediate risk prostate cancer. Late quality of life will be assessed with regular clinical exams and patient quality of life questionnaires.
Time Frame: Within 6 months of completion of radiation therapy
Population: as for outcome 1
Arm/Group | Focal SBRT With Intra-urethral Radiotransponder
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Each participant was assessed at baseline, during time of treatment, and during follow-up at 3, 6, 9, 12, 18, and 24 months after completion of treatment.
Arm/Group | Focal SBRT With Intra-urethral Radiotransponder
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
5 patients signed consent, 1 patient withdrew consent prior to start of treatment. The funding source informed they are no longer manufacturing radiotransponder. No similar product. Therefore, no longer proceeding with study and no data collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/34/NCT03458234/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT03458234/ICF_001.pdf